CLINICAL TRIAL: NCT06410170
Title: Correlation of Urinary and Serum Hormone Levels in Natural Cycle Frozen Embryo Transfer Cycles
Acronym: MIRA
Status: Not yet recruiting | Type: Observational
Sponsor: Ottawa Fertility Centre (Other)
Collaborators: Quanovate Tech Inc. (Industry)
Responsible Party: Principal Investigator, Dr. Jenna Gale, Research Director, Ottawa Fertility Centre
Other Study IDs: 2024-3364-17398-2
Record Dates: First submitted 2024-04-25; First posted 2024-05-13 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Fertility Issues
Keywords: Mira device; Fertility tracking; At home use
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Single Cohort Group: Evaluating the anticipated utility of the Mira device for detection of the LH surge, in natural cycle frozen embryo transfer protocols
  Interventions: Device: MIRA Device

INTERVENTIONS:
Device: MIRA Device — At home diagnostic testing
  Other Names: Device wands

SUMMARY:
To evaluate whether the measurement of urinary estrone glucuronide and luteinizing hormone (LH) concentrations with an at-home device is correlated with serum hormone levels within a natural cycle frozen embryo transfer protocol.

The hypothesis is that home urinary monitoring can reliably detect the LH surge and serve as a trigger for timing the FET. Results of this study may ultimately lead to change in clinical practice by reducing the number of clinic visits for serum monitoring, offering a more convenient, time and cost saving method of detection of LH surge. If the proposed protocol were feasible and widely accepted by patients, this would prompt the wide adoption of a less invasive but equally as effective FET protocol.

DETAILED DESCRIPTION:
A prospective multi-center cohort study evaluating the anticipated utility of the Mira device for detection of the LH surge, in natural cycle frozen embryo transfer protocols. All patients scheduled for undergoing natural cycle frozen embryo transfers at The Ottawa Fertility Centre (Ottawa, Ontario, Canada) and Olive Fertility Centre (Vancouver, British Columbia, Canada) with the ability to provide informed consent for participation will be eligible for inclusion. Each individual patient may only be included once in the study.

The objective of the proposed study is to evaluate whether the use of home urinary testing of quantitative estradiol metabolites and LH can be used to accurately predict ovulation and serve as a trigger for the gold standard of serum LH monitoring in a natural cycle protocol for frozen embryo transfer (FET). Its anticipated that this at home device will provide a reliable alternative to daily bloodwork, thereby reducing the number of daily visits for serum monitoring and also increased satisfaction and quality of life with the implementation of their use within these cycles.

Estrone glucuronide (E3G) and Pregnanediol-3-Glucoronide (PdG) are the major metabolites of estradiol (E2) and progesterone that can be measured in the urine. Similarly, LH is another hormone that is commonly measured during natural cycle FET cycles and can also be quantified in the urine. Urinary E3G, LH and PdG measurement are commercially available with an FDA and CE registered home device called the Mira Fertility Tracker ("Mira"). Correlation between the serum hormones and their respective urinary metabolites has been established but the efficacy of monitoring urinary E3G and LH has not been demonstrated in the context of natural cycle FET.

Therefore the study will take place within a true natural cycle protocol, whereby ovulation occurs spontaneously and is not triggered with exogenous hormones. Patients meet to discuss the approach to FET with their physician prior to proceeding with treatment. Patients are considered to be candidates for natural cycle protocol if they have regular menstrual cycles, ranging in length between 27-35 days and no luteal phase concern (i.e. significant luteal phase spotting, or evidence of a short luteal phase).

ELIGIBILITY:
Inclusion Criteria:

* All patients scheduled for a natural cycle frozen embryo transfer
* Agree to participate in the research study

Exclusion Criteria:

* There are no exclusions

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants that are presenting for a natural cycle frozen embryo transfer at The Ottawa and Olive Fertility Centre's
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
average delay in days | Through study completion, an average of 1 year
  delay in days of surge detection between the Mira device compared to the serum detection, corrected for the time of the tests.
Patient satisfaction Survey | Through study completion, an average of 1 year
  evaluate patient satisfaction with the use of the Mira device and willingness to utilize this device as an alternative to daily serum monitoring

SECONDARY OUTCOMES:
Progesterone metabolites | Through study completion, an average of 1 year
  Evaluate the proportion of cycles that have a rise in PdG (a urinary progesterone metabolite) prior to or at the time of their LH surge
BhCG urine vs Blood | Through study completion, an average of 1 year
  evaluate the correlation of urinary BhCG measurements relative to serum BhCG evaluation 12-14 days post embryo transfer.

CONTACTS AND LOCATIONS:
Overall Officials: Jenna Gale, MD, Principal Investigator — Ottawa Fertility Centre
Locations (1):
- Olive Fertility Centre, Vancouver, British Columbia, Canada